CLINICAL TRIAL: NCT04474782
Title: Analysis of Defocus Curve of Pre-Presbyopic and Emerging Presbyopic Patients
Status: Completed | Type: Observational
Sponsor: Vance Thompson Vision (Other)
Collaborators: Alcon Research (Industry)
Responsible Party: Sponsor
Other Study IDs: VT-2019-01
Record Dates: First submitted 2020-07-07; First posted 2020-07-17 (Actual); Last update posted 2021-03-30 (Actual); Status verified 2021-03

CONDITIONS: Presbyopia
MeSH Terms: conditions — Presbyopia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: There is not an intervention — There is not an intervention

SUMMARY:
Educating patients on visual performance with presbyopic correcting intraocular lenses is crucial. Understanding the defocus curve of pre-presbyopic and emerging presbyopic crystalline lens will provide eye care provides useful information to better educate patients on visual performance expectations after cataract surgery with a presbyopic correcting intraocular lens. Our objective will be to assess the subjective range of clear vision of a pre-presbyopic and emerging presbyopic patient population utilizing a defocus curve. A comparison of the pre-presbyopic and emerging presbyopic defocus curve to all FDA-approved presbyopic intraocular lenses will be discussed in the manuscript.

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to provide written informed consent on the IRB approved Informed Consent Form
2. 37-48 years of age
3. Phakic

Exclusion Criteria:

1. Previous cataract surgery
2. Any pathology for which, in the investigator's judgement, could reduce the subjects BCVA
3. Subjects that are unable to obtain 20/20 BCVA (i.e. amblyopia, etc.)

Ages: 37 Years to 48 Years | Sex: All
Age Groups: Adult
Study Population: A population of 30-60 subjects will be selected for testing. Subjects can be male or female, ages 37-48.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2019-10-17 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2020-08-31 (Actual)

PRIMARY OUTCOMES:
Change in LogMar visual acuity during vision testing on ETDRS with loose lenses | Screening/enrollment visit

CONTACTS AND LOCATIONS:
Locations (1):
- Vance Thompson Vision, Sioux Falls, South Dakota, United States

IPD SHARING:
Plan to Share IPD: No